CLINICAL TRIAL: NCT05908851
Title: Perioperative Pain Management for Total Shoulder Arthroplasty: A Pilot Non-Inferiority Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120986
Record Dates: First submitted 2023-04-25; First posted 2023-06-18 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Arthritis; Anesthesia, Local; Local Infiltration
MeSH Terms: interventions — Saline Solution; Ropivacaine; Morphine; Epinephrine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional Brachial Plexus Blockade (No Intervention): Ultrasound guided brachial plexus blocade with 10 ml of 0.5% ropivacaine using a high frequency linear array transducer.
- Local Infiltration Anesthesia (Experimental): High volume local infiltration anesthesia with 100 mL of 0.9% normal saline (57ml), 0.5% ropivacaine (40 ml), 10 mg morphine (10 mg/ml), 0.1 mg of epinephrine (0.1 mg/ml), and 30 mg of ketorolac (30 mg/ml) divided equally into a 20 ml five-zone field infiltration into the suprascapular notch/posterior capsule (suprascapular and axillary nerves), coracobrachialis muscle, anterior deltoid muscle, superior pectoralis major muscle, and skin incision at the conclusion of the procedure by the treating surgeon.
  Interventions: Drug: 100 mL of 0.9% normal saline (57ml), 0.5% ropivacaine (40 ml), 10 mg morphine (10 mg/ml), 0.1 mg of epinephrine (0.1 mg/ml), and 30 mg of ketorolac (30 mg/ml)

INTERVENTIONS:
Drug: 100 mL of 0.9% normal saline (57ml), 0.5% ropivacaine (40 ml), 10 mg morphine (10 mg/ml), 0.1 mg of epinephrine (0.1 mg/ml), and 30 mg of ketorolac (30 mg/ml) — Ultrasound guided brachial plexus blockade
  Other Names: High volume local infiltration anesthesia
  Arms: Local Infiltration Anesthesia

SUMMARY:
Total shoulder arthroplasty (TSA) is a common and effective treatment for end-stage shoulder pathologies. Over the past 25 years, implant designs have evolved and the indications for joint replacement have expanded significantly to include arthritis, rotator cuff arthropathy, complex shoulder trauma and trauma sequelae. This has resulted in a worldwide increase in rates of shoulder replacement surgery. The concomitant increased treatment burden for health care systems has prompted interest in strategies to improve the effectiveness and efficiency of patient care such as streamlining intraoperative procedures, mitigating complications, and reducing length of stay by providing outpatient surgical care. Outpatient lower extremity arthroplasty is commonplace and provides helpful information that can guide the development of outpatient TSA such as careful patient selection and the use of standardized perioperative pain management protocols. In lower extremity arthroplasty, several authors have described challenges associated with nerve blockade and the advantages of high-volume local infiltration analgesia (LIA) for outpatient arthroplasty. Proponents of outpatient TSA also describe the importance of patient selection, standardized perioperative protocols and implementation of comprehensive perioperative pain management strategies that can include the use of perioperative ultrasound guided interscalene brachial plexus blockade with a "single shot" injection, ultrasound guided interscalene brachial plexus blockade with a temporary indwelling catheter (ISB), LIA near the surgical site, and multimodal postoperative analgesics.

DETAILED DESCRIPTION:
A noninferiority clinical trial will be utilized for the study. Eighty patients undergoing primary TSA (anatomic or reverse TSA) with an orthopaedic surgeon at the Roth McFarlane Hand and Upper Limb Centre will be recruited into the study. The study participants (n=80) will be randomized preoperatively into either 1) the ultrasound guided ISB group (n=40) or 2) the high-volume LIA group (n=40). For the pilot study, the investigators will also measure recruitment rates, time to study completion, and drop-out rates.

All patients will undergo TSA through a standard deltopectoral approach. Postoperative rehabilitation will include routine protocols including sling protection for 6 weeks and the following progressive exercises: sling, pendulum, active-assisted range of motion, active range of motion, passive range of motion and shoulder girdle strengthening. Patients randomized to the ultrasound guided ISB group will receive brachial plexus blockade with 10 ml of 0.5% ropivacaine using a high frequency linear array transducer (Sonosite Edge II, FUJIFILM Sonsonite, Inc., Bothell, WA, USA). Patients randomized to the high-volume LIA group will receive 100 mL of 0.9% normal saline (57ml), 0.5% ropivacaine (40 ml), 10 mg morphine (10 mg/ml), 0.1 mg of epinephrine (0.1 mg/ml), and 30 mg of ketorolac (30 mg/ml) divided equally into a 20 ml five-zone field infiltration into the suprascapular notch/posterior capsule (suprascapular and axillary nerves), coracobrachialis muscle, anterior deltoid muscle, superior pectoralis major muscle, and skin incision at the conclusion of the procedure by the treating surgeon. Patients will be discharged with a standard prescription of multimodal analgesics including acetaminophen, ibuprofen, sustained release morphine, and short acting opioid.

In this case, because the LIA option is likely associated with lesser cost and lower risk of adverse events, non-inferior effectiveness for pain control would provide sufficient and clear evidence that the LIA is the preferred choice. The trial will follow CONSORT reporting guidelines . All measures will be administered though our Methods Centre web-based data collection and will be completed in clinic under the direction of a study coordinator. If a patient misses a follow-up, the web-based system will allow us to capture the outcome measures remotely. While investigators have selected multiple secondary outcome measures, they reflect important secondary dimensions and are measured with well-validated short forms that have low response burden. Potential mediators: Sex, age, gender-related pain expectations, occupation, and comorbid health status will be recorded as potential covariates. Sample size estimation: The criteria for sample size requirements for noninferiority trials is based on the smallest difference that is considered clinically relevant and the standard deviation expected from the sample. n=80 participants (n=40 per group) is a conservative estimate based on the ability to detect a moderate effect between study groups for a mean between-groups difference in the primary outcome .

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing total shoulder arthroplasty for:

* Osteoarthritis
* Rheumatoid arthritis
* Rotator cuff arthropathy
* Acute fracture
* Fracture sequelae.

Exclusion Criteria:

* Patients with known allergy to study medications
* Patients with obstructive sleep apnea
* Prior TSA
* patients previously on chronic narcotic medication
* patients who are unable to read English
* patients not able/willing to follow up for the study period of 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain VAS | 12 months
  Pain visual analogue scale - 10 point scale: 0 = no pain, 10 = worst pain imaginable.

SECONDARY OUTCOMES:
ASES Shoulder Score | 12 months
  ASES - Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
EQ5D | 12 months
  Patient Rated general health measure - 100 point scale: 0 = poor health, 100 = excellent health.
Shoulder Pain and Disability Index (SPADI) | 12 months
  Patient Rated Outcome: 0 - 130 rating scale - 0 = low pain and disability, 130 = high pain and disability.
Quick Disabilities of the Arm Shoulder and Hand: Q-DASH | 12 months
  Patient Rated Outcome: 100 point scale: 0 = disability, 100 = no disability
Western Ontario Osteoarthritis Shoulder Score (WOOS) | 12 months
  Patient Rated Outcome - 1900 point scale: 0 = excellent function, 1900 = poor function.
Constant Score | 12 months
  Patient Rated Outcome: 0 - 100 point rating scale: 0 = poor function, 100 = normal function
Single Assessment Numeric Evaluation: SANE Score | 12 months
  Patient Rated Outcome - 100 point rating scale: 0 = poor function, 100 = perfect function
Analgesia Diary | 3 months
  record of analgesics used

CONTACTS AND LOCATIONS:
Locations (1):
- St. Josephs Healthcare London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No